CLINICAL TRIAL: NCT01463852
Title: A Study of the Effect of Vinca Alkaloids on c-Jun N-terminal Kinase (JNK) Phosphorylation Status in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Study of the Effect of Vinca Alkaloids on c-Jun N-terminal Kinase (JNK) Phosphorylation in Patients With Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment underperformance.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D11199
Record Dates: First submitted 2011-10-31; First posted 2011-11-02 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: vincristine; JNK; phosphorylation; cll; vinca alkaloid; apoptosis
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell | interventions — Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vincrisitne 2mg (Experimental): Single Arm study: Vincristine 2mg administered IV by infusion over 5 minutes.
  Interventions: Drug: vincristine

INTERVENTIONS:
Drug: vincristine — Vincristine 2mg will be administered one time to participants. Blood samples will be collected pre and post dose.

SUMMARY:
In this proof-of-principle study, patients with chronic lymphocytic leukemia (CLL), who are scheduled to initiate treatment per the recommendations of their primary oncologist, will receive a single dose of vincristine 2 milligrams (mg). The objective is to determine if this single dose will induce rapid cell death in isolated CLL cells.

Vincristine 2 mg will be administered to the participants intravenously over 5 minutes. Blood samples will be collected from an intravenous line inserted into the contralateral limb to that where the vincristine was given, at time zero (pre-vincristine treatment), immediately after vincristine administration (within 2-10 minutes upon completion of administration) and at 1, 2, 4 and 6 hours post-vincristine treatment. Patients will then at a later date receive chemotherapy treatment as prescribed by their primary oncologist.

Within 7 days of vincristine administration, participants will receive a phone call from the research nurse to discuss potential toxicities. At the time of the initiation of standard chemotherapy treatment, the Principal Investigator will also meet with the participant to collect information regarding adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years old or older.
2. A diagnosis of Chronic Lymphocytic Leukemia(CLL) which is CD5/CD19/CD23 positive, confirmed by peripheral blood immunophenotyping and/or lymph node biopsy and immunophenotyping and/or bone marrow biopsy and immunophenotyping. CD23-negative CLL cases are eligible, however additional diagnostic confirmation should include absence of Cyclin D1 rearrangement [t(11;14)] as determined by standard laboratory methods (such as fluorescent in situ hybridization).
3. Patients are planning to start chemotherapy for CLL recommended and prescribed by their primary oncologist.
4. Peripheral blood lymphocyte count above 20,000/mm3
5. Be able to provide written informed consent

Exclusion Criteria

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients who are receiving any other investigational agents.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to vincristine.
4. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Liver function test abnormalities of ≥ grade 3 (total bilirubin >3 ULN (upper limit of normal), AST> 5 ULN, ALT> 5 ULN) as per CTCAE 4.0 criteria, or direct bilirubin ≥ 3.0 mg/dL
6. Pre-existing neuropathy grade 2 or greater as per CTCAE 4.0 criteria (moderate symptoms limiting instrumental activities of daily living - ADLs)
7. Patients who are pregnant or planning to become pregnant during their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
c-Jun N-terminal Kinase (JNK) activation | Change in JNK activation from baseline up to 6 hours post dose
  blood draws are collected pre-vincristine and at 10 minutes,1,2,4,and 6 hours post vincristine.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire, United States